CLINICAL TRIAL: NCT02053285
Title: Pilot Study of Dual-Energy Computed Tomography in Stage III Non-Small Cell Lung Cancer
Brief Title: Pilot Study of a Novel Type of CT Scan to Assess Treatment Response During Chemoradiotherapy for Stage III Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Dual-Energy Tomogr. | 12051502; 12051502 (Other: Rush University Medical Center)
Record Dates: First submitted 2014-01-23; First posted 2014-02-03 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dual-energy CT (DECT) provides information on the blood volume in tumors and lymph nodes. As tumors respond to treatment, preliminary data suggests that the blood volumes changes as well. Investigators are therefore using DECT to test whether it can be used on radiation treatment to rapidly assess response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged greater than 18 years with a diagnosis of stage III non-small cell lung cancer.
* Planned treatment with either definitive chemoradiotherapy or preoperative chemoradiotherapy followed by surgical resection.
* PET-CT study within 4 weeks of next available DECT study.
* Patients must have measurable primary and nodal disease, defined by at least one lesion (primary and lymph node) greater than 1 cm.
* Kidney function sufficient to tolerate iodine-based CT contrast.
* No allergy to iodine-based contrast.
* Ability to understand and the willingness to sign informed consent.

Exclusion Criteria:

* Participants with a prior history of thoracic radiotherapy.
* Participants may not be receiving any other study agents.
* Inability to tolerate CT contrast
* Pregnant women are excluded from this study because radiotherapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with radiotherapy, breastfeeding should be discontinued if the mother is treated with radiotherapy. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III lung cancer treated with chemoradiotherapy or chemoradiotherapy followed by surgery
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2019-05 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change in the tumor's maximum iodine related attenuation (IRA) from baseline to on-treatment DECT. | 0, 1, 3, 5
  This change in the maximum IRA will be compared with the change in the maximum standardized uptake value (SUV max) between baseline PET-CT and follow-up PET-CT at 3 months after treatment. For patients undergoing surgery, this change in the maximum IRA will be compared between patients who have a complete pathologic response, and those patients who do not.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Informed Consent Form (2015-05-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT02053285/ICF_000.pdf